CLINICAL TRIAL: NCT06707467
Title: Determination of the Effectiveness of Postural Exercises Combined With Occlusal Splint Therapy in Internal Temporomandibular Derangements
Brief Title: Evaluation of Postural Exercises in the Treatment of Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Berk Bilgen, PhD DDS Research Assistant, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-186
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Occlusal Splints; Temporomandibular Disorders (TMD)
Keywords: temporomandibular disorders; rocabado; occlusal splints; posture excercise
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Patients with internal temporomandibular derangement are divided into three groups. The first group receives only occlusal splint therapy. The second group undergoes occlusal splint therapy combined with Rocabado exercises, while the third group is treated with occlusal splint therapy combined with postural exercises. The effectiveness of the treatment protocols is evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nineteen patients with internal temporomandibular disarrangement-group 1 (Experimental): Nineteen randomly selected patients with internal temporomandibular disarrangement
  Interventions: Other: occlusal splints combined with rocabado exercise
- nineteen patients with internal temporomandibular disarrangement-group 2 (Active Comparator): nineteen randomly selected patients with internal temporomanidbular disarrangement
  Interventions: Other: occlusal splint
- nineteen patients with internal temporomandibular disarrangement-group 3 (Experimental): nineteen selected patients with internal temporomandibular disarrangements
  Interventions: Other: occlusal splint combined with posture exercise

INTERVENTIONS:
Other: occlusal splint — nineteen patients diagnosed with internal temporomandibular derangement will receive occlusal splint therapy, a treatment method with proven effectiveness.
  Arms: nineteen patients with internal temporomandibular disarrangement-group 2
Other: occlusal splints combined with rocabado exercise — Nineteen patients diagnosed with internal temporomandibular derangement will be provided with Rocabado exercises in addition to the proven-effective treatment method of occlusal splint therapy. This approach aims to evaluate whether Rocabado exercises have a positive effect on the treatment process.
  Arms: nineteen patients with internal temporomandibular disarrangement-group 1
Other: occlusal splint combined with posture exercise — Nineteen patients diagnosed with internal temporomandibular derangement will be provided with posture exercises in addition to the proven-effective treatment method of occlusal splint therapy. This approach aims to evaluate whether posture exercises have a positive effect on the treatment process.
  Arms: nineteen patients with internal temporomandibular disarrangement-group 3

SUMMARY:
Fifty-seven patients diagnosed with internal temporomandibular derangement will be included in the study and divided into three groups. All patients will be treated with a proven-effective occlusal splint. The first group will receive only occlusal splint therapy and will serve as the control group. The second group will receive occlusal splint therapy combined with Rocabado exercises, while the third group will receive occlusal splint therapy combined with postural exercises.

Before the treatment process, all patients will complete the Temporomandibular Disorders Diagnostic Criteria (TMD-DC) form. Pain intensity will be measured using the Visual Analog Scale (VAS), pain thresholds will be assessed using an algometer, and the following evaluations will be performed: Cervical Posture Assessment (Craniovertebral Angle with Goniometer)-Cervical Range of Motion Assessment (C-ROM)-Cervical Deep Flexor Muscle Endurance Test-Neck Disability Assessment (NDI - Neck Disability Index)-Psychiatric Assessment (HADS - Hospital Anxiety and Depression Scale).

After two months, patients will be recalled, and all tests will be repeated. The effectiveness of the three treatment protocols will then be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with internal temporomandibular disarrangement
* aged 18 years or older
* Willingness to participate in the study
* Ability to speak and understand Turkish, with no communication difficulties severe enough to impede understanding of the exercises

Exclusion Criteria:

* History of acute trauma in the TMJ or surrounding area
* TMJ dysfunction caused by a neurological condition
* History of surgical/invasive procedures or treatments on the TMJ
* Presence of infection or tumoral structures within intraoral structures
* History of tooth loss or use of dental prostheses
* History of surgical procedures in the cervical region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Investigation of the Effect of Postural Exercises and Rocabado Exercises on Pain Reduction | 2 months
  Three different treatment protocols will be applied to patients with internal temporomandibular derangement, and the results obtained after a 2-month treatment period will be compared to determine which method is the most effective. To evaluate treatment outcomes, the patients' pre- and post-treatment Visual Analog Scale (VAS) scores will be assessed, with a decrease in the mean VAS score indicating a reduction in pain. Additionally, the pain threshold in various facial regions will be measured with an algometer before and after treatment to identify which treatment protocol is more effective in reducing pain. By combining both outcomes, the most effective method for pain reduction will be determined.
Investigation of the Effect of Postural Exercises and Rocabado Exercises on Physiological Movements | 2 months
  Changes in cervical range of motion (C-ROM) and the craniovertebral angle will also be evaluated to determine the impact of the treatment methods on these parameters. In this way, the method that is more effective in improving physiological movements will be identified.

SECONDARY OUTCOMES:
Investigation of the Secondary Effects of Postural Exercises and Rocabado Exercises on Patient's Psychology | 2 months
  The effect of the treatment protocols applied to the three different groups on the general psychology of the patients will be measured using the Hospital Anxiety and Depression Scale (HADS). In this test, a higher score indicates a higher level of depressive symptoms, and a successful treatment is expected to result in a decrease in the test score.
Investigation of the Effect of Postural Exercises and Rocabado Exercises on the Mobility of the Neck and Jaw | 2 month
  The patient's neck movements will be assessed, and the range of jaw movements will be evaluated. The study aims to identify which treatment protocol leads to the most significant improvement in jaw and neck mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru K Mutlu, Clinical Prof., Study Director — Bandırma Onyedi Eylül University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)